CLINICAL TRIAL: NCT07271355
Title: Investigation of Mitomycin C PIPAC - FOLFIRI Combination for Unresectable Appendiceal or Colorectal Peritoneal Metastases Treatment (IMPACT): A Multicenter, Randomized, Open-Label, Phase 3 Trial
Brief Title: Pressurized Intraperitoneal Aerosolized Chemotherapy With Mitomycin for the Treatment of Unresectable Appendix or Colorectal Cancer With Peritoneal Metastases, The IMPACT Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24756; NCI-2025-08527 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24756 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-11-28; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Appendix Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Peritoneum; Stage IV Appendix Carcinoma AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (mitomycin PIPAC, FOLFIRI, bevacizumab) (Experimental): Patients receive mitomycin via PIPAC during on day 1 of each cycle. Cycles repeat every 6 weeks for 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after each mitomycin PIPAC treatment, patients receive FOLFIRI regimen, consisting of irinotecan IV over 90 minutes, leucovorin IV over 30 minutes, and fluorouracil IV over 46-48 hours on day 1 of each cycle (i.e., weeks 2, 4, 8, 10, 14, 16, etc). Cycles of FOLFIRI regimen repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after last cycle of mitomycin PIPAC, patients may also receive bevacizumab IV over 30-90 minutes at the discretion of the treating physician. Cycles of bevacizumab repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, collection of blood, ascites, and urine samples, as well as biopsies throughout the study. Patients may also undergo MRI during screening.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Questionnaire Administration
- Arm II (FOLFIRI, bevacizumab) (Active Comparator): Patients receive FOLFIRI regimen, consisting of irinotecan IV over 90 minutes on day 1 of each cycle, leucovorin IV over 30 minutes on day 1 of each cycle, and fluorouracil IV over 46-48 hours on day 1 of each cycle. Cycles repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after standard laparoscopy, patients also receive bevacizumab IV over 30-90 minutes on day 1 of each cycle. Cycles of bevacizumab repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may cross-over to Arm I (NOTE: Cross-over patients do not receive FOLFIRI regimen). Patients also undergo CT, collection of blood, ascites, and urine samples, as well as biopsies throughout the study. Patients may also undergo MRI during screening.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood, urine, and ascites
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given via PIPAC
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
  Arms: Arm I (mitomycin PIPAC, FOLFIRI, bevacizumab)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well pressurized intraperitoneal aerosolized chemotherapy (PIPAC) with mitomycin works versus (vs) standard chemotherapy (leucovorin calcium, fluorouracil, and irinotecan hydrochloride [FOLFIRI regimen] plus bevacizumab) in treating patients with appendix or colorectal cancer that cannot be removed by surgery (unresectable) and has spread from where it first started (primary site) to the abdominal cavity (peritoneal metastases). PIPAC is a new therapeutic approach that is minimally invasive, does not require surgery (laparotomy), and can be frequently repeated. Chemotherapy is delivered as a pressurized mist directly inside the abdominal cavity (peritoneum) during a minimally invasive surgery called a laparoscopy. The pressure helps the chemotherapy absorb into the cancer tissue and spread more evenly. Mitomycin is an antibiotic used as a chemotherapy drug. It stops or slows the growth of cancer cells and other rapidly growing cells by damaging their deoxyribonucleic acid (DNA). Standard chemotherapy drugs, such as those in the FOLFIRI regimen, are given via infusion into a vein (intravenously), and work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Another standard intravenous drug, bevacizumab, is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Giving mitomycin via PIPAC in combination with the standard FOLFIRI regimen, with or without bevacizumab, may work better than standard FOLFIRI plus bevacizumab alone in treating patients with unresectable appendix or colorectal cancer with peritoneal metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the overall survival of patients treated with mitomycin PIPAC (MMC-PIPAC) in combination with systemic FOLFIRI in comparison to those treated with systemic FOLFIRI/bevacizumab as a 2nd line therapy in patients with appendiceal or colorectal cancer with peritoneal metastases.

SECONDARY OBJECTIVES:

I. Compare progression-free survival between the two arms. II. Rate of completion of cytoreductive surgery.

III. Evaluate the Objective response rate by arm, assessed by:

IIIa. Peritoneal Regression Grading Score (PRGS) via histologic assessment of biopsies performed at each PIPAC cycle; IIIb. Laparoscopic Peritoneal Carcinomatosis Index (PCI) reduction; IIIc. Radiographic response by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1; IIId. Tumor marker (CEA) response rate. IV. Patient-reported health state/quality of life and symptoms before treatment, at 6 months and at 1-year, as measured by European Organisation for the Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC-QLQ30) and EORTC-Colorectal Cancer (CR29) for each arm.

EXPLORATORY OBJECTIVES:

I. Characterization of sub-clonal and tumor microenvironment evolution in response to therapy with a particular focus on immune and fibroblast subsets in the tumor and immune subsets in peripheral blood.

II. Correlating cell free DNA, ribonucleic acid (RNA), proteins and/or metabolites in blood and peritoneal fluid with burden of disease, survival and response to therapy.

III. Develop artificial intelligence and machine learning approaches for the characterization of peritoneal metastases by correlating video/photographic imaging features of peritoneal metastases to histologic features.

IV. Establish the feasibility of generating patient-derived xenografts, organoids, and cell lines from pre-treated colorectal and appendiceal cancer peritoneal metastases (City of Hope [COH] only).

V. Characterization of stool and tissue microbiome of patients on the study protocol.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive mitomycin via PIPAC during on day 1 of each cycle. Cycles repeat every 6 weeks for 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after each mitomycin PIPAC treatment, patients receive FOLFIRI regimen, consisting of irinotecan intravenously (IV) over 90 minutes on day 1 of each cycle, leucovorin IV over 30 minutes on day 1 of each cycle, and fluorouracil IV over 46-48 hours on day 1 of each cycle (i.e., weeks 2, 4, 8, 10, 14, 16, etc). Cycles of FOLFIRI regimen repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after last cycle of mitomycin PIPAC, patients may also receive bevacizumab IV over 30-90 minutes at the discretion of the treating physician. Cycles of bevacizumab repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive FOLFIRI regimen, consisting of irinotecan IV over 90 minutes on day 1 of each cycle, leucovorin IV over 30 minutes on day 1 of each cycle, and fluorouracil IV over 46-48 hours on day 1 of each cycle. Cycles repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after standard laparoscopy, patients also receive bevacizumab IV over 30-90 minutes on day 1 of each cycle. Cycles of bevacizumab repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may cross-over to Arm I (NOTE: Cross-over patients do not receive FOLFIRI regimen).

All patients also undergo computed tomography (CT), collection of blood, ascites, and urine samples, as well as biopsies throughout the study. Patients may also undergo magnetic resonance imaging (MRI) during screening.

After completion of study treatment, patients are followed up at 4 weeks and then every 8-12 weeks until death.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed appendiceal or colorectal cancer peritoneal metastases
* No extraperitoneal metastases except lung ≤ 5 lesions with largest ≤ 1cm as identified on CT imaging or MRI. CT scan or MRI to assess measurable disease must have been completed within 28 days prior to registration
* Visible peritoneal metastatic disease on cross-sectional imaging or diagnostic laparoscopy (does not have to be measurable by RECIST (v1.1)
* Completed at least 4 months (8 cycles) of first-line standard-of-care oxaliplatin-based systemic therapy without progression of disease. Or completed less than 4 months of oxaliplatin based therapy due to intolerance and without progressive disease. Or progressed on first-line standard-of-care oxaliplatin-based systemic therapy. Permissible first-line systemic therapies include leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) or capecitabine and oxaliplatin (XELOX) or fluorouracil, leucovorin, oxaliplatin and irinotecan (FOLFOXIRI). Receipt of anti-EGFR, anti-VEGF, or anti-BRAF therapy in the first-line is acceptable. Mismatch repair-deficient patients are permissible if they have progressed on first-line immunotherapy
* Not a candidate for cytoreductive surgery as determined by site investigator
* Fully recovered from the acute toxic effects of prior anti-cancer therapy to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or lower except alopecia, hearing loss, neuropathy, or non-clinically significant laboratory abnormalities
* Complete medical history and physical exam (To be performed within 28 days prior to Day 1 of protocol therapy)
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (To be performed within 28 days prior to Day 1 of protocol therapy)
* Platelets ≥ 100,000/mcL (To be performed within 28 days prior to Day 1 of protocol therapy)
* Hemoglobin ≥ 8 g/dL (To be performed within 28 days prior to Day 1 of protocol therapy)
* Serum albumin ≥ 2.8 g/dL (To be performed within 28 days prior to Day 1 of protocol therapy)
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease, then direct bilirubin < 1.5 mg/dL) (To be performed within 28 days prior to Day 1 of protocol therapy)
* Aspartate aminotransferase (AST) ≤ 5 x ULN (To be performed within 28 days prior to Day 1 of protocol therapy)
* Alanine aminotransferase (ALT) ≤ 5 x ULN (To be performed within 28 days prior to Day 1 of protocol therapy)
* Calculated creatinine clearance of ≥ 45 mL/min per 24-hour urine test or the Cockcroft-Gault formula (To be performed within 28 days prior to Day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test (To be performed within 28 days prior to Day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control (e.g. licensed hormonal/barrier methods or surgery intended to prevent pregnancy [or with a side effect of pregnancy prevention]) or abstain from heterosexual activity for the course of the study through at least 14 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* CROSS-OVER ARM INCLUSION: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* CROSS-OVER ARM INCLUSION: Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with Study PI approval
* CROSS-OVER ARM INCLUSION: Age: ≥ 18 years
* CROSS-OVER ARM INCLUSION: ECOG performance status of 0 or 1
* CROSS-OVER ARM INCLUSION: No extraperitoneal metastases except lung ≤ 5 lesions with largest ≤ 1cm as identified on CT imaging or MRI. CT scan or MRI to assess measurable disease must have been completed within 28 days prior to registration
* CROSS-OVER ARM INCLUSION: Progression on Control Arm of the Study as determined by RECIST v1.1. Non-radiographic progression will need to be assessed on a case-by-case basis by central review
* CROSS-OVER ARM INCLUSION: Fully recovered from the acute toxic effects of prior anti-cancer therapy to CTCAE grade 1 or lower except alopecia, hearing loss, neuropathy, or non-clinically significant laboratory abnormalities
* CROSS-OVER ARM INCLUSION: Complete medical history and physical exam (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: ANC ≥ 1,500/mcL (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Platelets ≥ 100,000/mcL (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Hemoglobin ≥ 8 g/dL (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Serum albumin ≥ 2.8 g/dL (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Total bilirubin ≤ 1.5 X ULN (unless has Gilbert's disease, then direct bilirubin <1.5 mg/dL) (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: AST ≤ 5 x ULN (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: ALT ≤ 5 x ULN (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Calculated creatinine clearance of ≥ 45 mL/min per 24-hour urine test or the Cockcroft-Gault formula (To be performed within 28 days prior to Day 1 of protocol therapy)
* CROSS-OVER ARM INCLUSION: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (To be performed within 28 days prior to Day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* CROSS-OVER ARM INCLUSION: Agreement by females and males of childbearing potential to use an effective method of birth control (e.g. licensed hormonal/barrier methods or surgery intended to prevent pregnancy [or with a side effect of pregnancy prevention]) or abstain from heterosexual activity for the course of the study through at least 14 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* More than 8 cycles of first line irinotecan therapy
* Progression on irinotecan
* Receipt of any second-line systemic chemotherapy (Note: Sequential administration of FOLFOX followed by FOLFIRI is considered second line therapy. However, FOLFOXIRI followed by FOLFIRI is considered first line as long as no more than 8 cycles of irinotecan are given)
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Strong CYP3A4 inducers/inhibitors within 14 days prior to Day 1 of protocol therapy
* Prior peritoneal-directed chemotherapy (Prior cytoreductive surgery is permitted)
* Participation in another clinical study with an investigational product administered in the last 2 months
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Low-grade appendiceal mucinous neoplasm or low-grade appendiceal mucinous adenocarcinoma
* Extraperitoneal metastases (except lung ≤ 5 lesions with largest being ≤ 1cm)
* Any history of bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy, or need for total parenteral nutrition. Even if the bowel obstruction resolved with conservative measures, the patient would be excluded. The exception is if the bowel obstruction was surgically addressed with ostomy, resection or bypass. This exception should be documented
* Fused mesenteric disease-causing mesenteric shortening and bowel sequestration ("cauliflowering")
* Bulky mesenteric disease where chemotherapy is unlikely to penetrate the tumor
* Contraindication to laparoscopy
* Rapid weight loss (> 10% in < 3 months)
* Ascites (> 2L drained per month)
* Adhesions involving > 50% of abdominal cavity on diagnostic laparoscopy
* Life expectancy < 6 months
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to Day 1 Cycle 1 of treatment

  * Patients receiving prophylactic antibiotics are eligible, provided the signs of active infection have resolved
* Any prior malignancy except adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for two years
* History of allergic or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to study agents (platinum-based compounds, etc.)
* History of allogeneic organ transplantation or other active primary immunodeficiency
* Active and uncontrolled infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), or human immunodeficiency virus (positive HIV 1/2 antibodies)
* Clinically significant uncontrolled illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase the risk of incurring AEs, or compromise the ability of the patient to give written informed consent
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* CROSS-OVER ARM EXCLUSION: Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* CROSS-OVER ARM EXCLUSION: Strong CYP3A4 inducers/inhibitors within 14 days prior to Day 1 of protocol therapy
* CROSS-OVER ARM EXCLUSION: Participation in another clinical study with an investigational product administered in the last 2 months other than the current study
* CROSS-OVER ARM EXCLUSION: Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* CROSS-OVER ARM EXCLUSION: Extraperitoneal metastases (except lung ≤ 5 lesions with largest being ≤ 1cm)
* CROSS-OVER ARM EXCLUSION: Any history of bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy, or need for total parenteral nutrition. Even if the bowel obstruction resolved with conservative measures, the patient would be excluded. The exception is if the bowel obstruction was surgically addressed with ostomy, resection or bypass. This exception should be documented
* CROSS-OVER ARM EXCLUSION: Fused or bulky mesenteric disease-causing mesenteric shortening and bowel sequestration
* CROSS-OVER ARM EXCLUSION: Contraindication to laparoscopy
* CROSS-OVER ARM EXCLUSION: Rapid weight loss (> 10% in < 3 months)
* CROSS-OVER ARM EXCLUSION: Ascites (> 2L drained per month)
* CROSS-OVER ARM EXCLUSION: Adhesions involving > 50% of abdominal cavity on diagnostic laparoscopy
* CROSS-OVER ARM EXCLUSION: Life expectancy < 6 months
* CROSS-OVER ARM EXCLUSION: Treatment with therapeutic oral or IV antibiotics within 14 days prior to Day 1 Cycle 1 of treatment

  * Patients receiving prophylactic antibiotics are eligible, provided the signs of active infection have resolved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 5 years
  The primary analysis will follow the intention-to-treat principle. OS will be summarized by the Kaplan-Meier method, and a one-sided stratified log-rank test will be used to compare treatment arms, with hazard ratios and 95 percent confidence intervals (CIs) estimated from Cox proportional hazards models.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to time of progression or death, whichever occurs first, assessed up to 5 years
  Progression is as assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 via contrast-enhanced computed tomography scan. CIs for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Win ratio | Up to 5 years
  Will be based on OS events being more clinically meaningful than PFS events.
Objective response rate | Up to 5 years
  Will be measured by RECIST 1.1, Peritoneal Regression Grading Score (PRGS), Peritoneal Carcinomatosis Index (PCI) on diagnostic laparoscopy, and biochemical response with serum tumor marker. For RECIST criteria, efficacy can be defined as the percentage of evaluable patients who have achieved complete response (CR), partial response (PR), or stable disease (SD). For PCI, efficacy can be defined as the percentage of evaluable patients who have achieved CR, PR, or SD. For PRGS, efficacy can be defined as the percentage of evaluable patients who have achieved a decrease in average PRGS over successive biopsies. The proportion of successes will be estimated by the number of successes divided by the total number of patients initiating therapy. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Incidence of post-operative surgical complications | Up to 4 weeks after final pressurized intraperitoneal aerosolized chemotherapy (PIPAC)
  Will be measured by Clavien-Dindo classification 4 weeks after each PIPAC. Results will be strictly descriptive in nature.
Rate of patients who have cytoreductive surgery | Up to 5 years
Patient-reported health state/quality of life and symptoms | Week 0 up to 12 months
  Will be measured by the European Organisation for the Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC-QLQ30) and EORTC-Colorectal Cancer (CR29). Patient-reported outcomes will be summarized with descriptive statistics.
Patient-reported number of good days | At 6 months and 1 year
  Patient-reported outcomes will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Raoof, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (5):
- United States (5):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - City of Hope at Chicago, Zion, Illinois